CLINICAL TRIAL: NCT01634633
Title: Endometrial Nerve Fibers Detection in Patients With Different Gynecological Pathologies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, reda mokhtar kamal ghanem, Mr, Ain Shams University
Other Study IDs: ENFD-25-2012; Ain shams maternity hospital (Other Grant/Funding Number: Ain shams maternity hospital)
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Gynecological Pathologies
Keywords: Endometrial nerve fibres

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to investigate the prevelence of endometrial nerve fibers in different gynecological pathologies

DETAILED DESCRIPTION:
The aim of this study is to investigate the prevelence of endometrial nerve fibers in different gynecological pathologies in addition to its relation to chronic pelvic pain

ELIGIBILITY:
Inclusion Criteria:

1. Age: 20-60 years of age.
2. Written and signed informed consent by the patient to participate in the study.
3. Women candidate for surgical intervention either via laparoscopy or laparotomy for different gynecological pathologies

Exclusion Criteria:

1. Suspected endometriosis.
2. Patient unwillingness to participate in the study.
3. No hormonal treatment for the last 6 months.
4. Suspected pregnancy.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The population of this study will be 300 patient undergoing laparoscopy or laparotomy for different gynecological diseases namely, polycystic ovarian disease (PCOD), ovarian cysts either benign or malignant, fibroid uterus, adenomyosis, endometrial hyperplasia and endometrial carcinoma
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-11 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Prevelencce of endometrial nerve fibers | 18 months
  Is to determine the prevelence of endometrial nerve fibers in different gynecological pathologies I via endometrial sampling

SECONDARY OUTCOMES:
Pelvic pain | 18 months
  Relating the density of endometrial nerve fibres to different types of pelvic pain

CONTACTS AND LOCATIONS:
Overall Officials: Reda MK Ghanem, M.B.B.Ch, Principal Investigator — Ain Shams University
Locations (1):
- Ain shams new maternity hospital, Cairo, Egypt